CLINICAL TRIAL: NCT01549327
Title: A Web-Based Person-Centred Navigation Tool for Newly Diagnosed Colorectal Cancer Patients: A Randomized Clinical Trial (RCT) to Assess Effects on Empowerment and Cost-Effectiveness (The TEN-C Study: Together to Enhance Navigation in Cancer)
Brief Title: The Effect of a Virtual Navigator on Colorectal Cancer Patient Empowerment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Carmen G. Loiselle, N., Ph.D., Associate Professor, Christine and Herschel Victor / Hope & Cope Chair in Psychosocial Oncology, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TEN-C; MOP 106710 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2012-02-29; First posted 2012-03-09 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Cancer
Keywords: Virtual Patient Navigation; Randomized Clinical Trial; Empowerment; Cost-Effectiveness; Cancer Information Preferences
MeSH Terms: conditions — Colorectal Neoplasms; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Care (Active Comparator): Participants who are randomized to the active comparator arm will receive routine care, which is the care routinely provided to the participant's patient population at the study centre.
  Interventions: Other: Routine Care
- Routine Care plus OIN (Experimental): OIN (Oncology Interactive Navigator) is the intervention. Participants who are randomized to routine care plus OIN will receive routine care and have unlimited access to the website for the study duration.
  Interventions: Other: Oncology Interactive Navigator

INTERVENTIONS:
Other: Oncology Interactive Navigator
  Arms: Routine Care plus OIN
Other: Routine Care
  Arms: Routine Care

SUMMARY:
For individuals diagnosed with colorectal cancer, exposure to up-to-date cancer information and support as well as guidance to access the most appropriate health care services is crucial for cancer self-management and support. Timely access to high quality cancer information is suggested to contribute to patient empowerment - defined as the perception of being better able to manage illness demands. With the advent of the information age, individuals are increasingly turning to online health information resources. The use of rigorous web-based tools is found to be an engaging and convenient way to access health information, while being tailored to people's needs and preferences. The present study seeks to examine the effects of a recently developed high quality and person-centred web-based tool, the Oncology Interactive Navigator (OIN) on patients' empowerment as well as document its cost-effectiveness. Participants newly diagnosed with colorectal cancer will be randomly assigned to experimental or control groups with the former having unrestricted access to the OIN for 8 months. Participants in the control group will receive care as usual. Information on background, medical characteristics, and empowerment will be collected as well as cost-effectiveness indicators. If producing the desired effects, the OIN could be proposed for national implementation across Canadian cancer centers. Work is currently underway to add over 23 types of cancer diagnosis to the OIN.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed, first diagnosis of colorectal cancer (all stages)
* within 20 weeks of when the individual was told s/he has colorectal cancer
* fluent in English or French; able and willing to complete questionnaires
* unrestricted home Internet access
* has used the Internet at least once in the past
* informed consent

Exclusion Criteria:

* previous history of CRC at any time, or any other cancer diagnosed within the last 5 years (exception: superficial skin cancer)
* medical or severe health problem
* terminal phase of colorectal cancer or too sick to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Empowerment | 8 months
  The main outcome for this trial is empowerment which is multidimensional. Key dimensions of empowerment are measured using five constructs from the health education impact Questionnaire system (reference). Repeated measures using analysis of variance will be used to compare patterns of change in empowerment constructs across time between trial groups.
  Reference:
  Osborne RH et al. Patient Educ Couns. 2007;66:192-201.

SECONDARY OUTCOMES:
Cost-effectiveness | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen G. Loiselle, N., Ph.D., Principal Investigator — McGill University
Locations (4):
- Canada (4):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Sunnybrook-Odette Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No